CLINICAL TRIAL: NCT07353853
Title: Pre-packaged Low-residue Diet for Bowel Preparation in Patients With Inflammatory Bowel Disease: A National Multicenter Randomized Controlled Non-inferiority Clinical Trial
Brief Title: Pre-packaged Low-residue Diet for Bowel Preparation in Patients With Inflammatory Bowel Disease
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Changhai Hospital (Other)
Responsible Party: Principal Investigator, Zhaoshen Li, professor, Changhai Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Diagnostic
Other Study IDs: CHEC2025-535
Record Dates: First submitted 2026-01-12; First posted 2026-01-21 (Actual); Last update posted 2026-01-21 (Actual); Status verified 2026-01

CONDITIONS: IBD (Inflammatory Bowel Disease); Colonoscopy; Colonoscopy: Bowel Preparation
Keywords: IBD; Colonoscopy; Bowel preparation
MeSH Terms: conditions — Inflammatory Bowel Diseases

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Nutrition Powder Group (Experimental): Participants will be provided with 6 sachets of pre-packaged low-residue diet one day prior to colonoscopy, to be consumed as needed in multiple servings during the day.Patients in this group will take a total of 2 liters of polyethylene glycol electrolyte solution for bowel preparation before colonoscopy, administered as split doses (1 L in the evening before and 1 L on the morning of the procedure).
  Interventions: Dietary Supplement: pre-packaged low-residue diet for bowel preparation
- Standard Low-Residue Diet Group (No Intervention): Participants follow standard low-residue diet guidelines (like ESPEN recommendations) for 24 hours before colonoscopy. This includes rice water, congee, noodles, and steamed eggs, while avoiding fruits/juices, vegetables, nuts, and other high-fiber foods.Patients in this group will take a total of 3 liters of polyethylene glycol electrolyte solution for bowel preparation before colonoscopy, administered as split doses (1 L in the evening before and 2 L on the morning of the procedure).

INTERVENTIONS:
Dietary Supplement: pre-packaged low-residue diet for bowel preparation — Participants will be provided with 6 sachets of pre-packaged low-residue diet one day prior to colonoscopy.Patients in this group will take a total of 2 liters of polyethylene glycol electrolyte solution for bowel preparation before colonoscopy.Stool specimens from patients will be sent for Genetic Analysis of gut microbiota.
  Arms: Nutrition Powder Group

SUMMARY:
The primary objectives of this project are twofold: firstly, to evaluate the role of Maifu Changqing® Complete Nutrition Formula Powder in bowel preparation for colonoscopy in patients with IBD; and secondly, to enhance the nutritional support and comfort of bowel preparation for IBD patients.

DETAILED DESCRIPTION:
The project workflow is divided into three main phases. During the project initiation phase, key tasks include designing the study protocol, developing the bowel preparation assessment questionnaire, and identifying collaborating centers. In the project implementation phase, we will conduct surveys on colonoscopy bowel preparation practices across participating centers, deliver training sessions, and collect the case report forms (CRF) for this project. During the conclusion phase, we will focus on evaluating the quality of the collected CRF data, striving to ensure its authenticity, comprehensiveness, and objectivity.

ELIGIBILITY:
Inclusion Criteria:

* Age: Adult patients between 18 and 75 years old;
* Diagnosis of IBD according to the 2023 Guidelines for the Diagnosis and Treatment of Inflammatory Bowel Disease;
* Voluntary participation in this clinical trial and provision of signed informed consent.

Exclusion Criteria:

* Patients with acute IBD, severe conditions, combined with major bleeding, suspected toxic megacolon, CD with severe intestinal stricture, gastrointestinal obstruction, or other conditions deemed unsuitable for colonoscopy by the physician;
* Patients with severe cardiac, pulmonary, hepatic, or renal dysfunction;
* History of previous colorectal surgical resection or use of medications that may affect intestinal motility within one week (e.g., antidepressants, sedatives, calcium channel blockers);
* History of stroke, spinal cord injury, or psychiatric disorders that impair compliance with bowel preparation and colonoscopy;
* Allergy to any component of the administered drugs or meal replacements;
* Pregnant or lactating women, and other individuals considered unsuitable for bowel preparation and colonoscopy by the physician.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1000 (Estimated)
Dates: Start 2026-01-01 (Actual); Primary Completion 2026-06-30 (Estimated); Study Completion 2026-06-30 (Estimated)

PRIMARY OUTCOMES:
Bowel preparation adequacy rate | 6 months
  Bowel preparation adequacy rate:Proportion of subjects with a Boston Bowel Preparation Scale (BBPS) score of ≥2 in each segment.The BBPS ranges from 0 to 3 per segment (total score 0-9), with higher scores indicating better bowel cleanliness.

SECONDARY OUTCOMES:
Subject Satisfaction | 6 months
  Subjects' subjective satisfaction with and willingness to repeat the entire bowel preparation process, assessed using a Visual Analogue Scale (VAS).The VAS is a 100-mm horizontal line anchored at "extremely dissatisfied" (0 mm) and "extremely satisfied" (100 mm). Higher scores indicate greater satisfaction.

CONTACTS AND LOCATIONS:
Overall Officials: Yu Bai, M.D., Principal Investigator — Changhai Hospital
Locations (1):
- Changhai Hospital, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: No